CLINICAL TRIAL: NCT03998293
Title: Direct Measurement of Proinsulin Clearance in Humans
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Newly available data suggests that measuring proinsulin clearance would not enhance predictive value of serum proinsulin
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Adrian Vella, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-003525; R01DK078645 (NIH)
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Healthy
MeSH Terms: interventions — Somatostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- proinsulin clearance (Other): all participants will be studied once where somatostatin will be used to block endogenous insulin secretion
  Interventions: Drug: Somatostatin

INTERVENTIONS:
Drug: Somatostatin — infused to block endogenous insulin secretion over a 4 hour period

SUMMARY:
Researchers are trying to determine how quickly proinsulin is cleared from the circulation.

DETAILED DESCRIPTION:
proinsulin clearance is necessary to determine the rate of secretion into the circulation

ELIGIBILITY:
Inclusion Criteria:

* Weight-stable, non-diabetic subjects from Biobank participants at Mayo Clinic, Rochester

Exclusion Criteria:

* Age < 25 or > 65 years (to avoid studying subjects who could have latent type 1 diabetes, or the effects of age extremes in subjects with normal or impaired fasting glucose).
* HbA1c ≥ 6.5%
* Use of glucose-lowering agents.
* For female subjects: positive pregnancy test at the time of enrollment or study
* History of prior upper abdominal surgery such as adjustable gastric banding, pyloroplasty and vagotomy.
* Active systemic illness or malignancy.
* Symptomatic macrovascular or microvascular disease.
* Hormone replacement therapy >0.625 mg premarin daily

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Proinsulin Clearance | through study completion, each study will take an average of 8 hours
  The half-life of proinsulin in a given individual
Proinsulin Distribution | through study completion, each study will take an average of 8 hours
  The volume of distribution of proinsulin in a given individual

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials